CLINICAL TRIAL: NCT00360555
Title: Best Tolerability: 50mg Twice Daily Versus 100 mg in the Evening Versus 25 mg Twice Daily Versus Placebo in Younger Women in North America
Brief Title: Uptitration Trial of Flibanserin Versus Placebo in Premenopausal Women With Hypoactive Sexual Desire Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 511.75
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- flibanserin (Experimental): flibanserin 25 mg b.i.d
  Interventions: Drug: flibanserin 50mg
- flibanserin 50mg (Experimental): flibanserin 50mg qhs/b.i.d
  Interventions: Drug: flibanserin 100mg
- flibanserin 100mg (Experimental): flibanserin 50mg b.i.d./100mg qhs
  Interventions: Drug: placebo
- placebo (Placebo Comparator): placebo comparator
  Interventions: Drug: flibanserin

INTERVENTIONS:
Drug: flibanserin — flibanserin 25 mg b.i.d
  Arms: placebo
Drug: flibanserin 50mg — flibanserin 50mg qhs/b.i.d.
  Arms: flibanserin
Drug: flibanserin 100mg — flibanserin 50 mg b.i.d/100mg qhs
  Arms: flibanserin 50mg
Drug: placebo — placebo comparator
  Arms: flibanserin 100mg

SUMMARY:
This trial is designed to assess the safety and efficacy of flibanserin in the treatment of premenopausal women with Hypoactive Sexual Desire Disorder (HSDD) that meets standard diagnostic criteria.

Efficacy for flibanserin will be assessed vs. a parallel placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are 18 years of age and older.
2. Premenopausal women having regular menstrual periods who have HSDD (decreased sexual desire), generalized acquired type, according to DSM IV-TR criteria.
3. Patient must meet minimum cut-off scores on questionnaires relating to sexual functioning and sexual distress.
4. Patients must be willing to try to have sexual activity (e.g., any act involving direct genital stimulation) at least once monthly.
5. Patients must be willing and able to use an electronic diary on a daily basis (e.g., have access to a working land line telephone for daily data transmissions).
6. At the Baseline Visit, patients must have complied with eDiary use adequately.
7. Patients must be in a stable, monogamous, heterosexual relationship that is secure and communicative, for at least 1 year prior to the Screen Visit. The partner is expected to be physically present at least 50% of each month.
8. Patients must have used a medically acceptable method of contraception for at least 3 months before the Baseline Visit (Visit 2) and continue to use that medically acceptable method of contraception during the trial.
9. In the investigators opinion, patients must be reliable, honest, compliant, and agree to co-operate with all trial evaluations as well as to be able to perform them.
10. Patients must be able and willing to give meaningful, written informed consent prior to participation in the trial, in accordance with regulatory requirements. Patients must have sufficient understanding to communicate effectively with the investigator, and be willing to discuss their sexual functioning with the investigative staff.
11. Patients must have a clinically acceptable Pap smear as read by a cytology facility (no evidence of malignancy or squamous intraepithelial lesions) within 6 months before the Screen Visit.
12. A score of 15 or higher on the FSDS-R at the screen Visit.

Exclusion Criteria:

1. Patients who have taken any medication noted in the protocols List of Prohibited Medications within 30 days before screening.
2. Patients whose sexual function was affected (enhanced or worsened) in the investigators opinion by any medication within 30 days before the Screen Visit and anytime prior to the Baseline Visit.
3. Patients with a history of drug dependence or abuse within the past one year.
4. Patients with a history of multiple severe reactions (i.e., allergic or oversensitivity to usual doses) to drugs that affect the brain.
5. Patients with a history of participation in a trial of another investigational medication within one month prior to the Screen Visit, or participation in any previous clinical trial of flibanserin.
6. Patients who meet accepted diagnostic criteria for sexual disorders that would interfere with improvement in HSDD (sexual aversion, substance-induced sexual problems, urge to live as a man, etc.
7. Patients who indicate that their sexual partner has inadequately treated sexual problems that could interfere with the patients response to treatment.
8. Patients who have entered the menopausal transition or menopause or have had a hysterectomy.
9. Patients with findings at the Screen Visit of infection, inflammation, undue tenderness, or shrinkage (atrophy) of the female organs.
10. Patients who are breast feeding or have breastfed within the last 6 months prior to the Baseline Visit.
11. Patients who are pregnant or have been pregnant within the last 6 months prior to the Baseline Visit.
12. Patients with a history of Major Depressive Disorder within 6 months prior the Screen Visit, a score indicating depression on a depression scale, a history of suicide attempt, or current suicidal ideation evident at the Screen or Baseline Visit.
13. Patients with a history of any other psychiatric disorders that could impact sexual function, risks patients safety, or may impact compliance.
14. Patients who have started psychotherapy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1584 (Actual)
Dates: Start 2006-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (77):
- United States (64):
  - 511.75.01015 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 511.75.01028 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 511.75.01051 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 511.75.01063 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 511.75.01017 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 511.75.01014 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 511.75.01042 Boehringer Ingelheim Investigational Site, Fair Oaks, California
  - 511.75.01022 Boehringer Ingelheim Investigational Site, Irvine, California
  - 511.75.01005 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 511.75.01053 Boehringer Ingelheim Investigational Site, Sacremento, California
  - 511.75.01045 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.75.01065 Boehringer Ingelheim Investigational Site, Aurora, Colorado
  - 511.75.01003 Boehringer Ingelheim Investigational Site, Englewood, Colorado
  - 511.75.01030 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 511.75.01066 Boehringer Ingelheim Investigational Site, Coral Gables, Florida
  - 511.75.01040 Boehringer Ingelheim Investigational Site, Fort Meyers, Florida
  - 511.75.01001 Boehringer Ingelheim Investigational Site, Gainesville, Florida
  - 511.75.01062 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 511.75.01032 Boehringer Ingelheim Investigational Site, Ocala, Florida
  - 511.75.01047 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 511.75.01073 Boehringer Ingelheim Investigational Site, Palm Bay, Florida
  - 511.75.01035 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 511.75.01010 Boehringer Ingelheim Investigational Site, South Miami, Florida
  - 511.75.01041 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 511.75.01033 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.75.01002 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 511.75.01006 Boehringer Ingelheim Investigational Site, Sandy Springs, Georgia
  - 511.75.01023 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.75.01031 Boehringer Ingelheim Investigational Site, Fort Wayne, Indiana
  - 511.75.01050 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 511.75.01043 Boehringer Ingelheim Investigational Site, Bingham Farms, Michigan
  - 511.75.01025 Boehringer Ingelheim Investigational Site, Chaska, Minnesota
  - 511.75.01024 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 511.75.01009 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 511.75.01060 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 511.75.01004 Boehringer Ingelheim Investigational Site, New Brunswick, New Jersey
  - 511.75.01037 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 511.75.01054 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 511.75.01069 Boehringer Ingelheim Investigational Site, Beachwood, Ohio
  - 511.75.01012 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.75.01071 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.75.01038 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 511.75.01048 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 511.75.01061 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.75.01020 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 511.75.01052 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 511.75.01059 Boehringer Ingelheim Investigational Site, Medfod, Oregon
  - 511.75.01021 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 511.75.01018 Boehringer Ingelheim Investigational Site, Jenkintown, Pennsylvania
  - 511.75.01067 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 511.75.01070 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 511.75.01064 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - 511.75.01049 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 511.75.01013 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 511.75.01027 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 511.75.01044 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 511.75.01011 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 511.75.01055 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.75.01068 Boehringer Ingelheim Investigational Site, Waco, Texas
  - 511.75.01007 Boehringer Ingelheim Investigational Site, Charlottesville, Virginia
  - 511.75.01057 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 511.75.01046 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.75.01019 Boehringer Ingelheim Investigational Site, Seattle, Washington
  - 511.75.01036 Boehringer Ingelheim Investigational Site, Middleton, Wisconsin
- Canada (13):
  - 511.75.02008 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 511.75.02002 Boehringer Ingelheim Investigational Site, North Vancouver, British Columbia
  - 511.75.02004 Boehringer Ingelheim Investigational Site, Woodstock, New Brunswick
  - 511.75.02005 Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 511.75.02010 Boehringer Ingelheim Investigational Site, Barrie, Ontario
  - 511.75.02011 Boehringer Ingelheim Investigational Site, London, Ontario
  - 511.75.02001 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 511.75.02007 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 511.75.02012 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 511.75.02014 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 511.75.02009 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 511.75.02013 Boehringer Ingelheim Investigational Site, Trois-Rivières, Quebec
  - 511.75.02003 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Thorp J, Simon J, Dattani D, Taylor L, Kimura T, Garcia M Jr, Lesko L, Pyke R; DAISY trial investigators. Treatment of hypoactive sexual desire disorder in premenopausal women: efficacy of flibanserin in the DAISY study. J Sex Med. 2012 Mar;9(3):793-804. doi: 10.1111/j.1743-6109.2011.02595.x. Epub 2012 Jan 12. PMID 22239862

RESULTS

PARTICIPANT FLOW:
Groups:
- Flibanserin 25 mg b.i.d: flibanserin: 25 mg twice daily
- Flibanserin 50mg Qhs/b.i.d: flibanserin: 50 mg once at bedtime/twice daily
- Flibanserin 50mg b.i.d./100mg Qhs: flibanserin: 50 mg twice daily/100 once at bedtime
- Placebo: flibanserin: placebo
Period: Overall Study
Arm/Group | Flibanserin 25 mg b.i.d | Flibanserin 50mg Qhs/b.i.d | Flibanserin 50mg b.i.d./100mg Qhs | Placebo
Started | 396 | 393 | 396 | 399
Completed | 274 | 259 | 251 | 287
Not Completed | 122 | 134 | 145 | 112

BASELINE CHARACTERISTICS:
Population: Demographic data are available for participants who were included in the "treated" analysis population of 1,581 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Flibanserin 25 mg b.i.d | Flibanserin 50mg Qhs/b.i.d | Flibanserin 50mg b.i.d./100mg Qhs | Placebo | Total
Number analyzed (Participants) | 396 | 392 | 395 | 398 | 1581
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 396 | 392 | 395 | 398 | 1581
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 396 | 392 | 395 | 398 | 1581
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 341 | 345 | 334 | 343 | 1363
  White Hispanic | 16 | 16 | 24 | 27 | 83
  Black Hispanic | 1 | 0 | 0 | 1 | 2
  Black | 33 | 27 | 29 | 21 | 110
  Asian | 5 | 4 | 8 | 6 | 23
  Asian Hispanic | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 346 | 344 | 349 | 352 | 1391
  Canada | 50 | 48 | 46 | 46 | 190

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Frequency of Satisfying Sexual Events (SSE) as Recorded in the eDiary.
Description: For endpoints collected on the eDiary, responses are accumulated on a monthly basis using the following algorithms.
  For satisfying sexual events:
  Total monthly events = 28 x (sum of the number of events) / (sum of number of days entered)
Time Frame: baseline to 28 weeks
Population: Participants who received at least one post-dose on-treatment efficacy assessment were included in the Full Analysis Set (FAS). Efficacy endpoints were analyzed primarily using the FAS.
Measure: Mean (Standard Deviation); unit: SSEs per 28 days
Arm/Group | Flibanserin 25 mg b.i.d | Flibanserin 50mg Qhs/b.i.d | Flibanserin 50mg b.i.d./100mg Qhs | Placebo
Number analyzed (Participants) | 376 | 369 | 371 | 381
SSEs per 28 days | 1.4 (3.5) | 1.4 (3.4) | 1.9 (5.3) | 1.1 (3.4)

2. Primary Outcome: Change From Baseline in the Monthly Sum of Responses Recorded in the eDiary to the Daily Desire Question.
Description: Change from baseline in the electronic diary (eDiary) Sexual Desire Monthly Total Score standardized to a 28-day period (score range 0-84). Change from baseline is calculated as the difference between the four week baseline period and Week 21 to Week 24. Patients were asked to record information daily in the eDiary throughout the trial. Every time the eDiary was completed, a desire question was asked. If a patient did not complete the diary on a given day, the patient was not asked to enter desire information for more than a 24-hour retrospective period. The desire item read "Indicate your most intense level of sexual desire in the last 24 hours / since your last visit." Potential responses included "no," "low," "moderate," or "strong" and was scored 0-3, with 0 indicating no desire and 3 indicating the highest level of desire:
  0 = No desire
  1. = Low desire
  2. = Moderate desire
  3. = Strong desire
Time Frame: baseline to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Flibanserin 25 mg b.i.d | Flibanserin 50mg Qhs/b.i.d | Flibanserin 50mg b.i.d./100mg Qhs | Placebo
Number analyzed (Participants) | 376 | 369 | 371 | 381
units on a scale | 7.9 (0.8) | 8.8 (0.8) | 8.5 (0.8) | 6.8 (0.8)

ADVERSE EVENTS:
Arm/Group | Flibanserin 25 mg b.i.d | Flibanserin 50mg Qhs/b.i.d | Flibanserin 50mg b.i.d./100mg Qhs | Placebo
Serious Adverse Events (participants affected / at risk) | 7/396 | 6/392 | 3/395 | 8/398
Other Adverse Events (participants affected / at risk) | 168/396 | 293/392 | 266/395 | 133/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 25 mg b.i.d (N=396) | Flibanserin 50mg Qhs/b.i.d (N=392) | Flibanserin 50mg b.i.d./100mg Qhs (N=395) | Placebo (N=398)
appendicitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitic acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrustion (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 25 mg b.i.d (N=396) | Flibanserin 50mg Qhs/b.i.d (N=392) | Flibanserin 50mg b.i.d./100mg Qhs (N=395) | Placebo (N=398)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 20 (25) | 25 (30) | 20 (21)
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 18 (20) | 16 (17) | 11 (13)
dizziness (Nervous system disorders) | 22 (23) | 54 (65) | 48 (54) | 8 (8)
somnolence (Nervous system disorders) | 29 (32) | 64 (73) | 47 (55) | 14 (14)
fatigue (General disorders) | 24 (25) | 60 (64) | 38 (40) | 27 (29)
nausea (Gastrointestinal disorders) | 20 (24) | 42 (51) | 47 (54) | 16 (18)
Headache (Nervous system disorders) | 29 (37) | 35 (65) | 45 (68) | 37 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No